CLINICAL TRIAL: NCT03720054
Title: An M-Health Intervention to Increase Activity Levels in Rural Veterans
Brief Title: An M-Health Intervention in Rural Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Philip Polgreen, Professor of Medicine, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201710866
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Veterans; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MapTrek (Experimental): Veterans in the intervention group receive a Fitbit and MapTrek, an interactive text-messaging platform. The only equipment needed is a Fitbit (we provide) and a smartphone (required prior to enrollment). Each week, veterans are assigned to a virtual walking route. Each day, they receive a text message with a link to the current route. The link will take them to a map where they can see their progress and the progress of others. A leaderboard provides information on how many steps each participant has taken. MapTrek also supports Street View on Google Maps, so veterans can explore what they would see if they were in that location. Throughout each race, patients will randomly receive challenge text messages. Completing a challenge awards bonus steps to propel their character along the map.
  Interventions: Behavioral: MapTrek
- Fitbit Only (Active Comparator): Veterans randomized to the control group will receive a Fitbit only. This will allow us to determine if changes in physical activity are due to MapTrek or simply by giving the veterans a Fitbit.
  Interventions: Behavioral: Fitbit

INTERVENTIONS:
Behavioral: MapTrek — Our objective is to report activity levels in our virtual environment to veterans, thereby encouraging them first, to walk more every day, and second, to maintain these new increased levels of physical activity. MapTrek will also motivate veterans to accumulate less sedentary time.
  Arms: MapTrek
Behavioral: Fitbit — Fitbit Only
  Arms: Fitbit Only

SUMMARY:
MapTrek is a mobile-phone-based web app that allows participants to take a virtual walk in interesting locations around the world while tracking their progress against the progress of other veterans on an interactive map. Steps are counted using a commercially available triaxial accelerometer (e.g. Fitbit), and users see their own updated progress overlaid on Google Maps, with Google Maps features (e.g. zooming, street view, etc.) available. The objective is to report activity levels in the virtual environment to veterans, thereby encouraging them first, to walk more every day, and second, to maintain these new increased levels of physical activity.

DETAILED DESCRIPTION:
All consented participants will be provided with a Fitbit and instructed to wear it all day for the next 9 weeks. This process should take approximately 15 to 45 minutes, depending on group assignment.

This, plus an exit survey and 3-month follow-up survey(given via text message or phone call, whichever the participant prefers), will be the extent of the participation in the control group.

Members of the intervention group will be instructed on how to use MapTrek, the virtual walking race. Data collected during the first week from the Fitbit will be used to compute baseline activity level. This baseline data will be used to place participants into an appropriate initial race group. Participants are placed into race groups with other individuals who are active at a similar level, so that groups will be competitive.

Each virtual walking race will begin on Monday and end on Sunday. Depending on each veteran's performance each week, group assignment may change. Participants will compete in 8 week-long races over the course of the study.

For each race, the participants will receive 2-4 text messages each day including a daily status report and a link to the current race. The participants will also periodically receive challenge text messages. If participants accept a challenge and meet it, they will be awarded bonus steps to help move them along the route in the race.

To win a race, participants must be the first to cross the finish line on the route for the week. There is a leaderboard within MapTrek that helps participants determine their standings within each race. Participants are allowed to choose a screen name to show on the leaderboard so that they may remain anonymous if desired.

For all participants, the investigators will collect first and last name and the last 4 digits of the participant's Social Security Number for consent documentation purposes and to look the person up in the VA medical record (CPRS). The following information will be collected from CPRS at baseline: age, sex, race, marital status, height, weight, body mass index, blood pressure, zip code, and current medications. Height, weight, body mass index, and blood pressure values will be collected again at the 9 week and 3 month follow ups. The following information will be collected from the MOVE! participation records at baseline: date enrolled in MOVE! program, number of MOVE! classes attended, weight when enrolled in the MOVE! program.

At the end of the 9 weeks of participation, participants will be contacted to complete an exit survey either via text message or phone call, whichever was stated as the preferred method at enrollment. This will take approximately 10 minutes to complete.

3 months after the study ends, the participants will be contacted to complete a 3-month follow-up survey either via text message or phone call, whichever was stated as the preferred method at enrollment. This will take approximately 10 minutes to complete.

Participants who do not respond will be contacted via text message and phone call up to 3 times. If participants still cannot be reached they will be considered lost to followup.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Be comfortable speaking and reading in English
* Have a BMI of at least 25
* Have a smartphone with texting and internet capabilities
* Be willing to download the Fitbit app onto their phone
* Must be a VA patient

Exclusion Criteria:

* Pregnancy
* Active mental health conditions that prevent them from providing own consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Self-Reported Ability to Participate | 9 weeks
  Ability (smartphone ownership, texting skill) to participate will be assessed via self-report from the participant.
Fitbit Usage | 9 weeks
  Amount of time (number of days, hours per day) spent wearing the Fitbit will be assessed.
Challenge Usage | 9 weeks
  Number of challenges participated in will be assessed.

SECONDARY OUTCOMES:
Total Number of Steps per Day | 9 weeks
  The Fitbit will provide the total number of steps that each veterans has taken per day.

OTHER OUTCOMES:
MapTrek Future Development Survey | 5 months
  Veterans will report areas of development within MapTrek to improve its future efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Health Care System, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No